CLINICAL TRIAL: NCT02071914
Title: A Randomised, Double-Blind, Placebo-Controlled, Single-Centre, Phase IIa Study in Healthy Volunteers to Evaluate the Efficacy and Safety of CT-P27 in an Influenza Challenge Model
Brief Title: A Study to Evaluate the Efficacy and Safety of CT-P27 in an Influenza Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P27 2.1
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Influenza A
Keywords: efficacy; safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CT-P27 10mg/kg (Experimental): CT-P27 will be administrated once in IV infusion.
  Interventions: Drug: CT-P27
- CT-P27 20mg/kg (Experimental): CT-P27 will be administrated once in IV infusion.
  Interventions: Drug: CT-P27
- Placebo (Placebo Comparator): Placebo will be administrated once in IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-P27 — Influenza A treatment drug.
  Arms: CT-P27 10mg/kg; CT-P27 20mg/kg
Drug: Placebo — Placebo.
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy of CT-P27 measured by quantitative PCR viral load from nasopharyngeal mucosa, compared to placebo.

DETAILED DESCRIPTION:
This study is a Randomised, Double-Blind, Placebo-Controlled, Single-Centre, Phase IIa study. All enrolled subjects will be given a single dose of 10 mg/kg CT-P27, 20 mg/kg CT-P27, or placebo intravenously and then followed by Day 36.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male & Female volunteers

Exclusion Criteria:

* Current clinically significant disease
* Pregnant or nursing mother
* Abnormal pulmonary function, nose or nasopharynx

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-02-15 (Actual); Primary Completion 2014-05-19 (Actual); Study Completion 2014-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SuEun Song, Study Director — Celltrion Inc.
Locations (1):
- Retroscreen Virology Ltd., London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P27 10mg/kg: CT-P27 will be administrated once in IV infusion.
  CT-P27 10 mg/kg: Influenza A treatment drug.
- CT-P27 20mg/kg: CT-P27 will be administrated once in IV infusion.
  CT-P27 20 mg/kg: Influenza A treatment drug.
- Placebo: Placebo will be administrated once in IV infusion.
  Placebos: Placebo.
Period: Overall Study
Arm/Group | CT-P27 10mg/kg | CT-P27 20mg/kg | Placebo
Started | 27 | 27 | 27
Completed | 27 | 27 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P27 10mg/kg | CT-P27 20mg/kg | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 27 | 81
Age, Continuous [Median (Full Range); unit: years] | 24.0 [20 to 39] | 25.0 [19 to 41] | 25.0 [18 to 42] | 25.0 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 12 | 32
  Male | 17 | 17 | 15 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - British | 22 | 23 | 18 | 63
  White - Irish | 0 | 1 | 0 | 1
  Any other white background | 5 | 2 | 4 | 11
  Asian or Asian British - Pakistani | 0 | 1 | 1 | 2
  Chinese | 0 | 0 | 1 | 1
  Any other Asian background | 0 | 0 | 2 | 2
  Any other mixed background | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Viral Load AUC (Day 1 to Day 9) by Nasopharyngeal Swab Quantitative PCR
Description: AUC of Viral Load, as Measured by Quantitative PCR of Nasopharyngeal Swab, Post-viral Challenge to the Last Assessment Day in Quarantine
Time Frame: Three times a day from Day 1(the day after virus inoculation) to Day 9
Population: The Infected Population included all subjects in the Efficacy Population who provided at least 2 positive nasopharyngeal swabs within 24 h when tested using quantitative PCR assay.
Measure: Mean (Standard Deviation); unit: Days*Eq log10 TCID50/mL
Arm/Group | CT-P27 10mg/kg | CT-P27 20mg/kg | Placebo
Number analyzed (Participants) | 20 | 20 | 21
Days*Eq log10 TCID50/mL | 6.474 (9.0090) | 6.974 (9.0817) | 11.639 (9.7982)

ADVERSE EVENTS:
Time Frame: up to Day 36/end-of-study (EOS) visit
Arm/Group | CT-P27 10mg/kg | CT-P27 20mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 4/27 | 3/27 | 7/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P27 10mg/kg (N=27) | CT-P27 20mg/kg (N=27) | Placebo (N=27)
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Infusion site pain (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Serious Adverse Events and Other (Not Including Serious) Adverse Events are treatment-emergent adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other